CLINICAL TRIAL: NCT04944992
Title: A Phase 2a, Randomized, Active-Comparator-Controlled, Open-Label Study to Evaluate the Efficacy and Safety of Efinopegdutide (MK-6024) in Individuals With Nonalcoholic Fatty Liver Disease
Brief Title: A Study of Efinopegdutide (MK-6024) in Participants With Nonalcoholic Fatty Liver Disease (NAFLD) (MK-6024-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6024-001; MK-6024-001 (Other: Merck); 2020-005136-30 (EudraCT Number)
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efinopegdutide (Experimental): Efinopegdutide 20 mg/mL administered by injection once weekly for 24 weeks in a dose-escalation regimen: 2.4 mg from day 1 to week 3, 5.0 mg from week 4 to 7, and 10.0 mg from week 8 to 24.
  Interventions: Drug: Efinopegdutide 20 mg/mL
- Semaglutide (Active Comparator): Semaglutide 1.34 mg/mL administered by injection once weekly for 24 weeks in a dose-escalation regimen: 0.25 mg from day 1 to week 3, 0.5 mg from week 4 to 7, and 1.0 mg from week 8 to 24.
  Interventions: Drug: Semaglutide 1.34 mg/mL

INTERVENTIONS:
Drug: Efinopegdutide 20 mg/mL — Subcutaneous injection in a dose-escalation administration of 2.4 mg, 5.0 mg, and 10.0 mg
  Other Names: MK-6024; HM12525A; JNJ-64565111
  Arms: Efinopegdutide
Drug: Semaglutide 1.34 mg/mL — Subcutaneous injection in a dose-escalation administration of 0.25 mg, 0.5 mg, and 1.0 mg
  Other Names: Ozempic®
  Arms: Semaglutide

SUMMARY:
The principal goal of this study is to determine the efficacy of efinopegdutide in liver fat reduction in participants with NAFLD. The primary hypotheses are that efinopegdutide is superior to semaglutide, or that efinopegdutide is superior to semaglutide by at least 10% with respect to mean relative reduction from baseline in liver fat content (LFC) after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* LFC ≥10% as assessed by MRI-PDFF at time of screening.
* Body Mass Index (BMI) ≥25 kg/m² and ≤50 kg/m² at time of screening.
* Stable weight (based on self-reporting) defined as ≤5% gain or loss of body weight for at least 3 months before screening visit.
* No history of Type 2 Diabetes Mellitus (T2DM) OR history of T2DM with an Glycated Hemoglobin (A1C) ≤8.5% at screening AND controlled by diet or a stable dose of metformin for the 3 months before screening.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP), or is a WOCBP and agrees to follow contraceptive guidance during the study intervention period and for at least 5 weeks after the last dose of study intervention.
* Participants in Taiwan are eligible between the ages of 20 to 70 years of age (inclusive).
* Participants in South Korea are eligible between the ages of 19 to 70 years of age (inclusive).

Exclusion Criteria:

* History of Type 1 Diabetes Mellitus (T1DM), diabetic ketoacidosis, or diabetes secondary to pancreatitis or pancreatectomy.
* Ongoing, inadequately controlled hypothyroidism or hyperthyroidism.
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasm type-2 syndrome.
* Recent event (within 6 months prior to screening) of congestive heart failure, unstable angina, myocardial infarction, arterial revascularization, stroke, or transient ischemic attack.
* History or evidence of chronic liver disease other than NAFLD or Non-Alcoholic SteatoHepatitis (NASH).
* Known history of cirrhosis.
* History of acute or chronic pancreatitis.
* History of a bariatric surgical procedure or a known clinically significant gastric emptying abnormality.
* History of malignancy ≤5 years prior to screening, except for skin cancer or cervical cancer.
* Clinically active hematologic disorder.
* Diagnosis of human immunodeficiency virus (HIV).
* Surgery requiring general anesthesia within 3 months before screening visit.
* History of organ transplantation, except for corneal transplant.
* Active diabetic proliferative retinopathy or a history of maculopathy.
* Untreated obstructive sleep apnea.
* History of treatment with any glucagon-like peptide-1 (GLP-1) receptor agonist within 6 months before screening.
* History of treatment with thiazolidinediones (ie, pioglitazone, rosiglitazone) within 6 months before screening.
* Previous use (within 3 months before screening) or current use of prescription weight-management medications or over-the-counter weight-loss medications or therapies.
* Treatment with systemic corticosteroid medication within 3 months before screening.
* Current treatment with anticoagulants (eg, warfarin, heparin).
* Inability to have an MRI-PDFF performed due to either severe claustrophobia, metallic implant that prevents MRI-PDFF examination, or any other contraindication to MRI-PDFF examination.
* Previous or current history of significant alcohol consumption (average of 7 standard drinks per week in females or 14 standard drinks per week in males) for a period of more than 3 consecutive months in the 24 months before screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (69):
- United States (9):
  - Catalina Research Institute, LLC ( Site 1939), Montclair, California
  - Sweet Hope Research Specialty, Inc ( Site 1902), Hialeah, Florida
  - Floridian Clinical Research, LLC ( Site 1950), Miami Lakes, Florida
  - Sensible Healthcare, LLC ( Site 1903), Ocoee, Florida
  - Lucas Research, Inc ( Site 1930), Morehead City, North Carolina
  - Texas Clinical Research Institute ( Site 1910), Arlington, Texas
  - Baylor College of Medicine-Advanced Liver Therapies ( Site 1960), Houston, Texas
  - American Research Corporation at Texas Liver Institute ( Site 1920), San Antonio, Texas
  - Clinical Trials of Texas, Inc. ( Site 1906), San Antonio, Texas
- Argentina (4):
  - CIPREC-Laboratorio ( Site 0104), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0101), Mar del Plata, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0105), Buenos Aires, Buenos Aires F.D.
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 0107), Buenos Aires
- Australia (2):
  - Westmead Hospital-Gastroenterology & Hepatology ( Site 0204), Westmead, New South Wales
  - Flinders Medical Centre-Hepatology and Liver Transplant Medicine ( Site 0201), Bedford Park, South Australia
- Heritage Medical Research Clinic ( Site 0302), Calgary, Alberta, Canada
- France (2):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital F-ENDOCRINOLOGY-DIABETOLOGY ( Site 0401), Dijon, Cote-d Or
  - centre hospitalier lyon sud-Endocrinologie, Diabète et Nutrition ( Site 0402), Pierre-Bénite, Rhone
- Israel (6):
  - Rambam Health Care Campus-Liver disease unit ( Site 0704), Haifa
  - Carmel Hospital-Liver Unit ( Site 0705), Haifa
  - Shaare Zedek Medical Center-Liver Unit ( Site 0703), Jerusalem
  - Rabin Medical Center ( Site 0701), Petah Tikva
  - Sheba Medical Center-The Liver Diseases Center ( Site 0700), Ramat Gan
  - Sourasky Medical Center-Gastroenterology and Liver Disease ( Site 0702), Tel Aviv
- Italy (5):
  - Policlinico Umberto I ( Site 0801), Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 0805), Milan, Lombardy
  - Humanitas-Medicina interna ed Epatologia ( Site 0800), Rozzano, Lombardy
  - Azienda Ospedaliero Universitaria ( Site 0803), Modena
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma-Medicine ( Site 0804), Verona
- Mexico (5):
  - Arké Estudios Clínicos S.A. de C.V.-Gastroenterology-Hepatology ( Site 0906), Mexico City, Mexico City
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 0908), Mexico City, Mexico City
  - Avix Investigación Clinica, S.C. ( Site 0907), Monterrey, Nuevo León
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan (, Mérida, Yucatán
  - Centro de Investigación y Gastroenterología ( Site 0902), Cuauhtémoc
- New Zealand (3):
  - Christchurch Hospital-Gastroenterology Research ( Site 1002), Christchurch, Canterbury
  - Auckland City Hospital-Liver Research Unit ( Site 1003), Auckland
  - Middlemore Clinical Trials ( Site 1000), Auckland
- Poland (4):
  - Nasz Lekarz Przychodnie Medyczne ( Site 1105), Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Warszawa ( Site 1107), Warsaw, Masovian Voivodeship
  - Clinical Medical Research ( Site 1101), Katowice, Silesian Voivodeship
  - ID Clinic ( Site 1100), Mysowice, Silesian Voivodeship
- Russia (4):
  - Center targetnoy therapy ( Site 1203), Moscow, Moscow
  - New Technologies of Medicine Clinic ( Site 1204), Dzerzhinskiy, Moscow Oblast
  - Saint Petersburg City Polyclinic 117-endocrinology department ( Site 1201), Saint Petersburg, Sankt-Peterburg
  - Astarta Clinic ( Site 1202), Saint Petersburg, Sankt-Peterburg
- South Korea (5):
  - Soon Chun Hyang University Bucheon Hospital ( Site 1304), Bucheon-si, Kyonggi-do
  - Inha University Hospital-Gastroenterolgy/Hepatology ( Site 1303), Incheon
  - Severance Hospital, Yonsei University Health System ( Site 1305), Seoul
  - Samsung Medical Center-Gastroenterology/Internal Medicine ( Site 1302), Seoul
  - Korea University Guro Hospital ( Site 1300), Seoul
- Spain (5):
  - Hospital Universitario Virgen de la Victoria-UGC Endocrinologia y nutricion ( Site 1405), Málaga, Andalusia
  - CHUS - Hospital Clinico Universitario ( Site 1403), Santiago de Compostela, La Coruna
  - Hospital Universitari Vall d'Hebron-Liver Unit - Department of Internal Medicine ( Site 1400), Barcelona
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA-Gastroenterologia y Hepatologia ( Site 1402), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Unidad de Ensayos Clínicos de Aparato Digestivo ( Site 1404), Seville
- Taiwan (3):
  - NATIONAL CHENG-KUNG UNI. HOSP.-Liver Research team of National Cheng Kung University Hospital ( Site, Tainan
  - National Taiwan University Hospital ( Site 1501), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Division of hepatology, department of gastroenterology (, Taoyuan District
- Turkey (Türkiye) (6):
  - Dokuz Eylül Üniversitesi-Endocrinology and Met. ( Site 1610), Balçova, İzmir
  - Ankara University Department of Hematology, Clinical Research Unit ( Site 1603), Ankara
  - Hacettepe Universitesi-internal diseases ( Site 1602), Ankara
  - Gazi Universitesi-gastroenterology ( Site 1605), Ankara
  - Bezmialem Vakf Üniversitesi-Gastroenterology ( Site 1606), Istanbul
  - Istanbul University Capa Campus-Gastroenterology ( Site 1604), Istanbul
- Ukraine (5):
  - Ukrainian Research Institute of Therapy ( Site 1704), Kharkiv, Kharkivs’ka Oblast’
  - L.T. Mala National Institute of Therapy of NAMS of Ukraine-Department of Aging Studies and Prevent, Kharkiv, Kharkivs’ka Oblast’
  - Poltova Oblast Clinical Hospital IM.M.V.Sklifosovskoho ( Site 1710), Poltava, Poltava Oblast
  - Communal Non-profit Enterprise "City Hospital #6" of Zaporizhzhia City Council-Therapy department (, Zaporizhia, Zaporizhzhia Oblast
  - Adonis Plus-Outpatient department ( Site 1701), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Romero-Gomez M, Lawitz E, Shankar RR, Chaudhri E, Liu J, Lam RLH, Kaufman KD, Engel SS; MK-6024 P001 Study Group. A phase IIa active-comparator-controlled study to evaluate the efficacy and safety of efinopegdutide in patients with non-alcoholic fatty liver disease. J Hepatol. 2023 Oct;79(4):888-897. doi: 10.1016/j.jhep.2023.05.013. Epub 2023 Jun 22. PMID 37355043
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 51 clinical sites in 16 countries.
Pre-assignment Details: Participant flow as per the database cutoff date of 19OCT2022.
Period: Overall Study
Arm/Group | Efinopegdutide | Semaglutide
Started | 72 | 73
Completed | 64 | 71
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efinopegdutide | Semaglutide | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (11.0) | 50.7 (10.9) | 49.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 33 | 32 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 26 | 51
  Not Hispanic or Latino | 46 | 47 | 93
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 62 | 63 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/M^2] | 35.2 (5.7) | 33.5 (5.0) | 34.3 (5.4)
Weight [Mean (Standard Deviation); unit: kg] | 100.2 (18.9) | 94.4 (18.9) | 97.3 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Relative Reduction From Baseline in Liver Fat Content (LFC) Measured by Magnetic Resonance Imaging-Estimated Proton Density Fat Fraction (MRI-PDFF), Evaluated by Blinded Independent Central Review (BICR) After 24 Weeks
Description: LFC was measured with liver images taken by MRI-PDFF and analyzed by BICR. Relative Reduction from Baseline to Week 24 = (Baseline - Week 24) / Baseline x 100%. Mean relative reduction from baseline in liver fat content is presented.
Time Frame: Baseline and up to ~24 Weeks
Population: All randomized participants who had received at least 1 injection (including only partial) of study intervention and had at least 1 assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Reduction
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Reduction | 72.7 [66.8 to 78.7] | 42.3 [36.5 to 48.1]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least squared means = 30.4, 90% CI 2-sided [22.1 to 38.7]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an adverse event is presented.
Time Frame: Up to ~29 weeks
Population: All randomized participants who received at least 1 injection (including only partial) of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percentage of Participants | 88.9 | 72.6
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; difference in percentage = 16.3, 95% CI [3.5 to 29.1]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study intervention due to adverse event is presented.
Time Frame: Up to ~24 weeks
Population: All randomized participants who received at least 1 injection (including only partial) of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percentage of Participants | 5.6 | 0
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in percentage = 5.6, 95% CI [0.4 to 13.5]

4. Secondary Outcome: Mean Absolute Reduction From Baseline in LFC Measured by MRI-PDFF (Evaluated by BICR) After 24 Weeks
Description: LFC was measured by liver images taken by MRI-PDFF and analyzed by BICR. The absolute reduction from baseline to Week 24 = Baseline - Week 24. The mean absolute reduction from baseline in LFC after 24 weeks of treatment is presented.
Time Frame: Baseline and up to ~24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of liver fat
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percentage of liver fat | 14.9 [13.6 to 16.3] | 8.8 [7.5 to 10.1]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in least squared means = 6.1, 90% CI 2-sided [4.6 to 7.7]

5. Secondary Outcome: Mean Percent Change From Baseline in Body Weight After 24 Weeks
Description: Body weight in kilograms was measured using a standardized, digital scale. The mean percent change from baseline in body weight after 24 weeks is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -8.5 [-9.5 to -7.5] | -7.1 [-8.1 to -6.2]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Superiority; p = 0.085, Mixed Models Analysis; Difference in Least Squared Means = -1.4, 90% CI 2-sided [-2.7 to -0.1]

6. Secondary Outcome: Mean Percent Change From Baseline in Total Cholesterol After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in total cholesterol. The mean percent change in total cholesterol is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -15.2 [-18.2 to -12.2] | -8.0 [-11.0 to -5.0]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in Least Squared Means = -7.2, 90% CI 2-sided [-11.2 to -3.1]

7. Secondary Outcome: Mean Percent Change From Baseline in Non-High Density Lipoprotein-Cholesterol (Non-HDL-C) After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in non-HDL-C. The mean percent change in non-HDL-C is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -16.8 [-20.5 to -13.0] | -11.0 [-14.8 to -7.3]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in least squared means = -5.7, 90% CI [-10.9 to -0.6]

8. Secondary Outcome: Mean Percent Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C) After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in HDL-C. Mean percent change in HDL-C is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -8.1 [-11.2 to -5.1] | 3.6 [0.6 to 6.6]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in least squared means = -11.7, 90% CI [-15.8 to -7.7]

9. Secondary Outcome: Mean Percent Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in LDL-C. The mean percent change in LDL-C is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -13.0 [-17.4 to -8.6] | -6.9 [-11.3 to -2.6]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in least squared means = -6.1, 90% CI [-12.0 to -0.1]

10. Secondary Outcome: Mean Percent Change From Baseline in Triglycerides (TG) After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in triglycerides. The mean percent change in triglycerides is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -30.9 [-35.6 to -25.8] | -23.3 [-28.5 to -17.7]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in least squared means = -7.6, 90% CI 2-sided [-14.3 to -0.9]

11. Secondary Outcome: Mean Percent Change From Baseline in Apolipoprotein B (apoB) After 24 Weeks
Description: Fasting blood samples were collected at baseline and after 24 weeks of treatment to assess mean percent change in apoB. The mean percent change in apoB is presented.
Time Frame: Baseline and up to ~24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Efinopegdutide | Semaglutide
Number analyzed (Participants) | 72 | 73
Percent Change | -14.7 [-18.2 to -11.1] | -9.2 [-12.8 to -5.7]
Statistical Analysis 1: Comparison: Efinopegdutide vs Semaglutide; Test type: Other — Difference (Efinopegdutide - Semaglutide) in %; Difference in least squared means = -5.4, 90% CI 2-sided [-10.4 to -0.4]

ADVERSE EVENTS:
Time Frame: Death and adverse events up to ~29 weeks
Description: Every participant is counted a single time for each applicable non-serious adverse event. A specific non-serious adverse event appears on this report only if its incidence in one or more of the columns is greater than the percent incidence specified in the report title, prior to rounding. A system organ class appears on this report only if one or more specific non-serious adverse events in that system organ class occurred during the study period.
Arm/Group | Efinopegdutide | Semaglutide
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/73
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/73
Other Adverse Events (participants affected / at risk) | 57/72 | 44/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efinopegdutide (N=72) | Semaglutide (N=73)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efinopegdutide (N=72) | Semaglutide (N=73)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 9 (15) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 7 (10) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (16) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (32) | 13 (29)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 5 (5)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 5 (6)
Nausea (Gastrointestinal disorders) | 20 (38) | 23 (36)
Vomiting (Gastrointestinal disorders) | 12 (23) | 11 (12)
Fatigue (General disorders) | 1 (1) | 6 (6)
COVID-19 (Infections and infestations) | 8 (8) | 10 (10)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Lipase increased (Investigations) | 4 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 11 (13)
Dizziness (Nervous system disorders) | 4 (7) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT04944992/Prot_SAP_000.pdf